CLINICAL TRIAL: NCT06746519
Title: A Phase I/II , Multicenter, Open Label Clinical Study Evaluating the Safety, Pharmacokinetics, and Efficacy of the Combination of the Menin Inhibitor BN104 for the Treatment of Patients With Acute Myeloid Leukemia
Brief Title: BN104 in Combination With Chemotherapy or Targeted Agents for Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chen Suning (Other)
Collaborators: BioNova Pharmaceuticals (Shanghai) LTD. (Industry)
Responsible Party: Sponsor-Investigator, Chen Suning, Principal Investigator, The First Affiliated Hospital of Soochow University
Organization: The First Affiliated Hospital of Soochow University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BN104-105
Record Dates: First submitted 2024-12-03; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BN104 Combined Intensive Chemotherapy in patients with newly diagnosed AML (Experimental)
  Interventions: Drug: BN104 combined Intensive Chemotherapy or Venetoclax/Azacitidine
- BN104 Combined Venetoclax/Azacitidine in patients with newly diagnosed AML (Experimental)
  Interventions: Drug: BN104 combined Intensive Chemotherapy or Venetoclax/Azacitidine
- BN104 Combined Venetoclax/Azacitidine in patients with relapsed/refractory AML (Experimental)
  Interventions: Drug: BN104 combined Intensive Chemotherapy or Venetoclax/Azacitidine

INTERVENTIONS:
Drug: BN104 combined Intensive Chemotherapy or Venetoclax/Azacitidine — The starting dose cohort(200mg BID N104) combined Intensive Chemotherapyor Venetoclax/Azacitidine. Each treatment cycle is anticipated to be 28 days in length, although cycle delays may be made due to delayed count recovery.

SUMMARY:
The Phase I/II trial is to learn the safety, pharmacokinetics, and preliminary efficacy of BN104 taken twice daily combined with Intensive Chemotherapy or Venetoclax/Azacitidine in patients with acute myeloblastic leukemia.

DETAILED DESCRIPTION:
The study is divided into 2 phases. Phase1 dose escalation part will enroll 90 patients to evaluate safety and tolerance of BN104 taken twice daily combined with Intensive Chemotherapy or Venetoclax/Azacitidine in patients with newly diagnosed or relapsed/refractory (R/R) acute myeloblastic leukemia with specific mutations (KMT2A gene rearrangement ,NPM1 gene mutation and NUP98 rearrangement). Patients will be allocated into 3 cohorts based on their disease status quo. Each cohort will use 3+3 dose escalation model, the starting dose level is 200mg of BN104 taken twice daily combined with Intensive Chemotherapy or Venetoclax/Azacitidine.

- Cohort A: Newly diagnosed AML patients with specific mutations who are suitable to receive BN104 combined with intensive chemotherapy(cytarabine with idarubicin or daunorubicin), which short as"7+3 induction regimen", consisting of remisson introdcution,consolidation and BN104 maintenance phase. Patients who achieve a complete remission (CR), complete remission with partial hematologic recovery (CRh), or complete remission with incomplete hematologic recovery (CRi) after 1 or 2 induction cycles may proceed on to consolidation therapy. Patients who do not achieve CR,CRh or CRi after 1 or 2 induction regimens will be considered a treatment failure and thus will be terminated from study treatment. Patients entering the consolidation phase then received an intravenous infusion of cytarabine 1-2 g/m2 every 12 hours (Q12H), using a total of 6 doses, which could be administered either consecutively at D1-3 or separately at D1, D3, and D5, depending on the study center's treatment routine. In each treatment cycle, the indicated dose of BN104 was given orally twice daily until the next cycle of consolidation treatment. Patients entering the consolidation phase receive at least 1 cycle of consolidation therapy and a maximum of 4 cycles.

After completion of consolidation therapy, patients who remain in CR, CRh, or CRi may continue to receive BN104 monotherapy maintenance therapy at the indicated dose administered twice daily for 1 cycle every 28 days until completion of 26 cycles of maintenance therapy, disease relapse/progression, receipt of hematopoietic stem cell transplantation, intolerable toxicity, loss to visit, withdrawal of informed consent, death, or other circumstances that, in the judgment of the investigator, require the termination of study drug, whichever occurs first.

* Cohort B: Newly diagnosed AML patients with specific mutations who are ≥75 years of age or <75 years of age but are not suitable for intensive chemotherapy due to co-morbidities. The regimen is BN104 taken twice daily combined with azacitidine and venetolax. Venetolax (100 mg, day 1; 200 mg, day 2; 400 mg, days 3-28) orally in combination with azacitidine 75 mg/(m2-d) subcutaneously x 7 days (D1-7), and after the target administered dose of Venegra was reached, BN104 was administered orally at the indicated dose twice daily in a continuous manner (D1-28, cycle 1 as D4-28) in 28-day treatment cycles.
* Cohort C: relapsed/refractory AML patients with specific mutations, prior treatment failure with menin inhibitors is required. The regimen is BN104 taken twice daily combined with azacitidine and venetolax.

Any patient may receive HSCT after termination of study treatment at any stage if assessed by the investigator to be amenable to hematopoietic stem cell transplantation (HSCT.) Patients whose patients are still in CR, CRh, or CRi after receiving HSCT may still continue to initiate BN104 monotherapy if they meet the appropriate criteria.

Phase II expansion part will enroll 30-45 patients and be conducted at the selected dose level to further evaluate the safety and tolerability of BN104 combined with Intensive Chemotherapy or Venetoclax/Azacitidine, as well as preliminary efficacy in Acute leukemia subjects with specific mutations (KMT2A gene rearrangement, NPM1 gene mutation and NUP98 mutation).

* Cohort D: Newly diagnosed AML patients with KMT2A rearrangements, NPM1 mutations, or NUP98 rearrangements who are fit for intensive chemotherapy.
* Cohort E: Newly diagnosed AML patients with KMT2A rearrangements, NPM1 mutations or NUP98 rearrangements who are unfit for intensive chemotherapy.
* Cohort F: relapsed/refractory AML patients with KMT2A rearrangement, NPM1 mutation or NUP98 rearrangement.

It is planned to enroll 10-15 patients in each cohort accordingly

ELIGIBILITY:
Inclusion Criteria:

* Have been fully informed about the study and have voluntarily signed the ICF;
* Patients with newly diagnosed primary AML according to the 2022 World Health Organization (WHO) criteria (Groups A and B) or patients with relapsed/refractory AML who have been previously treated with menin inhibitor monotherapy (Group C) and have an intermediate or poor prognosis according to the 2022 ELN Risk Stratification, as well as a defined combination of NPM1 mutation or NUP98 rearrangement or KMT2A rearrangement
* Peripheral blood leukocyte count ≤ 25 x 109/L (limited to patients enrolled in groups B and C, where hydroxyurea is allowed to control peripheral blood leukocyte count)
* Aged 18 years or older;
* ECOG (GroupA and B:0,1,2; GroupC:0,1,2,3)
* For patients in group B, unfit for intensive chemotherapy is defined as:≥75 years of age or;Age ≥18 years and age <75 years with any of the following co-morbidities;ECOG score of 2 or 3;Cardiac history: congestive heart failure requiring treatment, or ejection fraction ≤50%, or chronic stable angina;DLCO ≤ 65% or FEV1 ≤ 65%;Creatinine clearance ≥30 ml/min and <45 ml/min;Liver injury total bilirubin > 1.5 x ULN but ≤ 3 x ULN.
* For patients in group C, previous failed treatment with menin inhibitors is required;
* adequate hepatic, renal, and cardiac function, as defined:Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal range (ULN);Total bilirubin ≤ 1.5 x ULN* and in patients with Gilbert disease, total bilirubin ≤ 3 x ULN;Creatinine clearance ≥ 45 ml/min* as estimated by the Cockcroft-Gault formula (if <45 ml/min, enrollment is allowed if creatinine ≤ 130 µmol/L); Left ventricular ejection fraction ≥ 45%*; Note: In Phase II studies, ALT or AST may be relaxed to ≤5 x ULN if the investigator assesses that the elevated ALT or AST is due to leukemia invasion of the liver;For patients <75 years of age enrolled in Group B, total bilirubin ≤ 3 × ULN, creatinine clearance ≥ 30 ml/min, or left ventricular ejection fraction < 50% are allowed;
* for patients with D-dimer test result > 5×ULN in the screening period, relevant tests (e.g. review of coagulation function after a certain time interval, ultrasound of deep veins of the lower limbs, etc.) are required to exclude deep vein thrombosis, hypercoagulable state of blood and disseminated intravascular coagulation before enrollment;
* expected survival of more than 12 weeks as judged by the investigator;
* Be willing to attend study visits as required by the study protocol
* female patients of childbearing potential or male patients whose female partners are of childbearing potential must agree to use an effective method of contraception, such as a double-barrier method of contraception, condoms, oral or injectable contraceptives, and intrauterine devices (IUDs), for the duration of the study and within 30 days of the last study dose. Postmenopausal women (>45 years of age and menopause of more than 1 year) and surgically sterilized women are exempt from this condition.

Exclusion Criteria:

* have active central nervous system (CNS) leukemia;
* a known history of clinically significant liver disease, including viral or other hepatitis or cirrhosis:Positive hepatitis B surface antigen (HBsAg) serology requires a negative hepatitis B virus (HBV) DNA test for enrollment; For patients with hepatitis C virus (HCV) antibody serology positive, a negative HCV RNA test result is required for enrollment.
* known human immunodeficiency virus (HIV) infection;
* pregnant (positive screening pregnancy test) or lactating females;
* meet any of the following cardiac-related criteria:Hereditary long QT interval syndrome or QTcF > 450 msec;Various clinically significant cardiovascular diseases, including acute myocardial infarction, unstable angina pectoris, coronary artery bypass grafting within 6 months prior to enrollment, congestive heart failure graded by the New York Heart Association (NYHA) as grade 2 or higher (inclusive);
* the patient has suffered from other malignant tumors within the past 5 years, except for radically treated basal cell carcinoma of the skin, carcinoma in situ of the breast or carcinoma in situ of the cervix;
* have received prior anti-leukemia therapy (for patients in Groups A and B), except for the following: use of hydroxyurea or leukocyte monocloning for control of white blood cell count, or treatment with all-trans retinoic acid due to initial suspicion of acute promyelocytic leukemia, or use of nondemethylating medications for the treatment of MDS
* for patients in Group C, prior anti-leukemia therapy, including chemotherapy, radiotherapy, hormonal therapy, targeted therapy, or immunotherapy, administered less than 2 weeks or 5 half-lives (whichever is shorter) prior to the start of study treatment; for patients who have undergone autologous hematopoietic stem cell transplantation or CAR-T therapy within 60 days prior to the start of study treatment, or have not recovered from toxicity associated with ASCT or CAR-T therapy Exclusion will be required for those who have had an allogeneic HSCT within 100 days prior to the start of study treatment, or if the patient still has a combination of active acute and chronic graft-versus-host disease, or if the patient still requires immunosuppressive therapy;
* pre-existing treatment with targeted menin (for Group A and B patients)
* pre-existing non-hematologic toxicities that have not returned to grade 0 or 1 (except alopecia areata);
* patients who have had a chest CT within 1 month prior to screening and suggestive of pulmonary nodules need to undergo T-SPOT (T-cell spotting test for tuberculosis infection) during the screening period, and those with positive results need to be excluded (no additional tests are required if no chest CT has been performed within 1 month prior to screening);
* uncontrolled active infection:Patients with non-serious infectious complications (e.g., oral Candida infection or uncomplicated urinary tract infection, etc.) for which oral/topical anti-infective therapy is being applied may be enrolled;Patients with severe infections requiring hospitalization or intravenous antibiotic therapy within 14 days prior to enrollment, patients with no evidence of infection, and patients receiving prophylactic anti-infective, antifungal, or antiviral therapy for prolonged neutropenia may be enrolled;Patients treated with intravenous antibiotics or hospitalized for febrile neutropenia, but no evidence of infectious etiology is found, and patients with a normal temperature for more than 72 hours without antipyretic medication may be enrolled;
* patients with known dysphagia, short bowel syndrome, gastroparesis, or other conditions that limit oral drug intake or gastrointestinal absorption;
* patients with a history of severe allergy to menin inhibitors or hypersensitivity to any component of BN104
* inadequate patient compliance with participation in this clinical study as judged by the investigator
* any other disease, metabolic abnormality, physical examination abnormality, or clinically significant laboratory test abnormality that, in the judgment of the investigator, gives reason to suspect that the patient has a disease or condition that is inappropriate for the use of the study medication, or that will interfere with the interpretation of the results of the study, or that places the patient at high risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2024-12-25 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of BN104 in combination with Venetoclax/Azacitidine or intensive chemotherapy | At the end of Cycle1 (Cycle1 Day28)
  Incidence of DLTs (evaluated at the end of cycle 1 for each dose level);

SECONDARY OUTCOMES:
Peak concentration (Cmax) | At the first Cycle, and Day1 of Cycle 2 (each cycle is 28days)
  Assess the Cmax of BN104 and its metabolite BNM-1263
Auc(0-last） | At the first Cycle, and Day1 of Cycle 2 (each cycle is 28days)
  Assess the area under the plasma concentration-time curve from time zero to the last quantifiable time point of BN104 and its metabolite BNM-1263
CR | At the screening, Cycle1Day28, Cvcle4Day1, Cycle7Day1, Cycle10Day1 (do the efficacy assessment each 3 cycles, each cycle is 28 days)
  To evaluate the CR rate of BN104 in combination with Venetoclax/Azacitidine or intensive chemotherapy
ORR (CR+CRh+CRi+PR+MLFS) | At the screening, Cycle1Day28, Cycle4Day1, Cycle7Day1, Cycle10Day1 (do the efficacy assessment each 3 cycles, each cycle is 28 days)
  To evaluate the ORR rate of BN104 in combination with Venetoclax/Azacitidine or intensive chemotherapy
DOR | At the screening, Cycle1Day28, Cycle4Day1, Cycle7Day1, Cycle10Day1 (do the efficacy assessment each 3 cycles, each cycle is 28 days)
  To evaluate the DOR of BN104 in combination with Venetoclax/Azacitidine or intensive chemotherapy
EFS | At the screening, Cycle1Day28, Cycle4Day1, Cycle7Day1, Cycle10Day1 (do the efficacy assessment each 3 cycles, each cycle is 28 days)
  To evaluate the EFS of BN104 in combination with Venetoclax/Azacitidine or intensive chemotherapy
RFS | At the screening, Cycle1Day28, Cycle4Day1, Cycle7Day1, Cycle10Day1 (do the efficacy assessment each 3 cycles, each cycle is 28 days)
  To evaluate the RFS of BN104 in combination with Venetoclax/Azacitidine or intensive chemotherapy
OS | At the screening, Cycle1Day28, Cycle4Day1, Cycle7Day1, Cycle10Day1 (do the efficacy assessment each 3 cycles, each cycle is 28 days)
  To evaluate the OS of BN104 in combination with Venetoclax/Azacitidine or intensive chemotherapy

OTHER OUTCOMES:
MRD negativity rate | At the screening, Cycle1Day28, Cycle4Day1, Cycle7Day1, Cycle10Day1 (do the efficacy assessment each 3 cycles, each cycle is 28 days)
  Assessment of CR with minimal residual disease (MRD) negativity and CRc with MRD negativity rate of BN104 in combination with Venetoclax/Azacitidine or intensive chemotherapy in patients with relapsed/refractory AML harboring specific gene alterations.
PD: MEIS1 | At the screening and the end of Cycle 1 (each cycle is 28 days)
  Assessment of the effect of BN104 in combination with intensive chemotherapy or Venetoclax/Azacitidine on MEIS1
PD: HOXA9 | At the screening and the end of Cycle 1 (each cycle is 28 days)
  Assessment of the effect of BN104 in combination with intensive chemotherapy or Venetoclax/Azacitidine on HOXA9

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China